CLINICAL TRIAL: NCT04257500
Title: Does Vaginal Delivery of Combined Hormonal Contraception Affect the Risk of Metabolic Syndrome in Overweight/Obese Women With PCOS
Acronym: RING-PCOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Andrea Roe, MD, MPH (Other)
Responsible Party: Sponsor-Investigator, Andrea Roe, MD, MPH, Assistant Professor of Obstetrics and Gynecology, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 834422
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — etonogestrel; NuvaRing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Contraceptive Ring (Experimental): Etonogestrel/ethinyl estradiol vaginal ring (NuvaRing), which releases 120 mcg of etonogestrel and 15 mcg of ethinyl estradiol daily.
  Interventions: Drug: Etonogestrel/ethinyl estradiol vaginal ring

INTERVENTIONS:
Drug: Etonogestrel/ethinyl estradiol vaginal ring — 16 weeks of continuous use of contraceptive vaginal ring
  Other Names: NuvaRing

SUMMARY:
A prospective study to determine the metabolic effects of the contraceptive vaginal ring among overweight and obese women with polycystic ovary syndrome (PCOS). We will recruit a total of 40 participants and study use of the vaginal ring over a 4-month period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS according to Rotterdam criteria, with at least 2 of 3 of the following criteria: oligomenorrhea (≤8 periods per year), clinical or biochemical hyperandrogenism, and polycystic ovaries on ultrasound
* Body mass index ≥25 and ≤45 kg/m2
* In good general health according to the investigators' discretion
* Willing to avoid pregnancy for the duration of the study

Exclusion Criteria:

* Current pregnancy or desire for pregnancy during course of study
* Current breastfeeding
* Second-trimester pregnancy within four weeks prior to initiation of NuvaRing or third-trimester pregnancy within 6 months prior to initiation of NuvaRing
* Use of hormonal contraception within four weeks prior to initiation of NuvaRing
* Diagnosis of metabolic syndrome. Metabolic syndrome will be defined according to the updated Adult Treatment Panel III as 3 or more of the following criteria: blood pressure ≥130/85 mm Hg, waist circumference >35 inches, fasting glucose ≥110 mg/dL, TG ≥150 mg/dL, HDL-C <50 mg/dL.
* Contraindications to NuvaRing use:

  * Age ≥ 35 plus tobacco use
  * Current or past deep vein thrombosis or pulmonary embolism
  * Cerebrovascular disease
  * Coronary artery disease
  * Thrombogenic valvular or rhythm diseases of the heart (such as subacute bacterial endocarditis with valvular disease or atrial fibrillation)
  * Inherited or acquired coagulopathy
  * Headaches with focal neurological symptoms or migraine headaches with aura
  * Age ≥ 35 plus any migraine headaches
  * Liver tumors, benign or malignant
  * Undiagnosed abnormal uterine bleeding
  * Current or past breast cancer or other estrogen- or progestin-sensitive cancer
  * Hypersensitivity to any of the components of NuvaRing
  * Use of hepatitis C drug combinations containing ombitasvir/paritaprevir/ritonavir
* Medical comorbidities:

  * 21-hydroxylase deficiency, congenital adrenal hyperplasia
  * Untreated thyroid disease
  * Untreated hyperprolactinemia
  * Type 1 or 2 diabetes mellitus
  * Uncontrolled liver disease
  * Uncontrolled renal disease
  * Current alcohol abuse
  * Hypertension ≥ 140 mm Hg average systolic or ≥ 90 mm Hg average diastolic in women using anti-hypertensive medication
  * Hypertension ≥ 150 mm Hg average systolic or ≥ 100 mm Hg average diastolic in women not using anti-hypertensive medication
  * History of or current gynecologic cancer
  * Triglycerides >=250 mg/dL
  * Current use of lipid-lowering or weight loss agents
  * Participation in any study of an investigational drug or device or biologic agent within 30 days
  * Suspected adrenal or ovarian tumor secreting androgens
  * Suspected Cushing's syndrome
  * Bariatric surgery within 12 months
  * Other medical concerns that in the judgment of the investigator may compromise safety of the participant or confound the reliability of compliance and information acquired in this study

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-03 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
Incidence of Metabolic Syndrome | 4 months
  Metabolic Syndrome defined according to the updated Adult Treatment Panel III as 3 or more of the following criteria: blood pressure ≥130/85 mm Hg, waist circumference >35 inches, fasting glucose ≥110 mg/dL, TG ≥150 mg/dL, HDL-C <50 mg/dL.

SECONDARY OUTCOMES:
Change in low-density lipoprotein (LDL) measure | 4 months
Change in high-density lipoprotein (HDL) measure | 4 months
Change in triglycerides measure | 4 months
Change in apolipoprotein A | 4 months
Change in apolipoprotein B | 4 months
Change in advanced lipid testing measure | 4 months
Change in cholesterol efflux capacity | 4 months
Change in fasting insulin level | 4 months
Change in fasting 2 hour oral Glucose Tolerance Test result | 4 months
Change in Testosterone | 4 months
Change in Ferriman-Gallwey Hirsutism score | 4 months
  A lower score indicates less hirsutism. The F-G scoring system has a minimum value of 0, and a maximum value of 36.
Body Mass Index | 4 months
Change in scoring on the Center for Epidemiologic Studies Depression Scale | 4 months
  The range of values is zero to 60, with the higher scores indicating the presence of more depressive symptoms.
Change in scoring on the State-Trait Anxiety Inventory | 4 months
  The State-Trait Anxiety Inventory measures both state and trait anxiety, the scores range from 20 to 80, with higher scores correlating with greater anxiety.
Change in scoring on Polycystic Ovary Syndrome Quality of Life Questionnaire | 4 months
  Worse quality of life is associated with a lower score on the questionnaire, with a range score from 30 to 210.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Roe, MD MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States